CLINICAL TRIAL: NCT06792994
Title: A Prospective Observational Trial to Assess Treatment Sequences and Factors That Impact Overall Sur-vival in Patients With Chronic Lymphocytic Leukaemia (CLL) Treated Within First-line Studies of the GCLLSG
Acronym: CLL2000
Status: Not yet recruiting | Type: Observational
Sponsor: German CLL Study Group (Other)
Collaborators: GELLC (Grupo Español de Leucemia Linfocítica Crónica) (Other); Nordic Lymphoma Group (Network); Polish Adult Leukemia Group (Other); HOVON - Dutch Haemato-Oncology Association (Other)
Responsible Party: Sponsor
Other Study IDs: CLL2000
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Long-term observation, CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Optional: Additional blood samples taken no more than once a year as part of routine care (no additional venous puncture is required).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patienst with CLL who received at least firstline treatment within a clinical trial: This trial will enroll patients who received first-line treatment in either CLL13, CLL14, or CLL17 trial. On ground of feasibility the sample size of the study is estimated at approximately 1800-2100 patients in total. No formal sample size calculation has been performed
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — The data of this observational trial will be collected as part of routine patient care. Data relating to the time period between the end of participation in the clini-cal first-line trial (CLL13, CLL14, or CLL17) and inclusion in the observational trial will be documented retrospectively at the time point of inclusion in the observa-tional trial. From inclusion in the observational trial, data on survival, long-term efficacy, quality of life, and safety will be collected prospectively

SUMMARY:
This observational trial is designed to investigate long-term survival with regard to the primary endpoint overall survival (OS) after start of first-line treatment.

DETAILED DESCRIPTION:
Primary objective:

To assess the overall survival (OS) from initiation of first-line treatment in patients who received different first-line therapies within the CLL13, CLL14, or CLL17 clinical trials.

Rationale for primary objective:

CLL is the most common leukaemia in adults in the western countries with an age-standardized incidence between 4 and 5 cases per 100,000 person-years and about 5,500 new CLL cases in Germany1. The clinical course of CLL is highly variable and can be predicted by clinical staging (according to Rai and Binet2,3) as well as genetic4, serum and other markers. Due to the increasing effectiveness of approved first-line therapies, some patients with CLL experience a normal life expectancy. Therefore, the total duration of clinical trials would need to be enormously extended in order to capture data on OS which is operationally not practicable. Moreover, a number of effective treatment options are available for follow-up therapies. Hence, the analysis of OS might not only be affected by the choice of first-line therapy but also by subsequent therapies and other competing factors that should be collected. Studies on long-term survival of patients with CLL have primarily relied on registry data5 and population-based studies6 and were conducted outside of clinical trials. These studies only occasionally consider specific comorbidities7,8, are retrospective in nature9, and often have limited observation periods. In addition, a potential accrual bias may be difficult to address within the format of registry data collection.

Prospective follow-up of patients would enable more comprehensive analyses within a predefined study patient population. This observational trial aims to prospectively analyze OS for a predefined study population. Patients who received first-line treatment in CLL1310, CLL1411, or CLL17 trials conducted by the German CLL Study group (GCLLSG) will be included to carry out this comprehensive analysis of OS in a well-defined patient population. To capture OS, all data that could influence OS, including but not limited to the presence of genomic risk factors and concomitant conditions at different time points, age, sex, country, subsequent lines of therapy and the occurrence of other diseases including causes of death, will also be recorded. In addition, data that had been collected within the initial first-line studies will be included in the analyses.

Secondary objectives:

To assess efficacy, measured by different time-to-event parameters from second-line treatment, and additionally from first-line treatment, particularly for those patients who have not yet received subsequent treatment lines.

Quality of life and safety (types, frequencies and follow-up adjusted incidence rates of second primary malignancies [SPM] and Richter's transformations [RT] as well as causes of death) will be assessed.

Rationale for secondary objectives:

OS and quality of life are considered the two most important endpoints in clinical research (Leary A. et al. Viewpoint Lancet 2024 ). Hence, with prolonged survival times and competing causes of death it is rather difficult to adequately capture these endpoints.

Patients with CLL have a significantly higher risk of developing SPMs compared to the general population12-16. The underlying mechanisms for this increased risk are not fully understood, but likely involve a combination of factors including tumor microenvironment, immunosuppression17, genetic predisposition, previous treatment15,18, aging and environmental exposures19. These SPMs can include various types of skin cancers such as non-melanoma skin cancer and malignant melanoma, as well as solid tumors (e.g., lung, breast, colon) and other hematologic malignancies (e.g., acute myeloid leukemia, non-Hodgkin lymphoma). With improved efficacy of treatment options with targeted agents, there is growing recognition, that the increased risk of SPMs may influence the OS of patients with CLL. The collection of long-term data based on the choice of first-line treatment in CLL patients and numbers, type and duration of subsequent therapies is essential not only for the analysis of OS, but equally for understanding the frequency of RT/SPMs. Such data will support informed treatment decision-making, risk stratification, and personalized medicine approaches, ultimately improving patient outcomes and guiding the development of safer and more effective CLL therapies. Therefore, investments in longitudinal data collection and collaborative research initiatives focusing on this important aspect of CLL management are warranted to optimize patient care and advance our understanding of CLL treatment-related complications.

In addition, progression-free survival (PFS) and time-to-next CLL treatment (TTNT) in patients who underwent their initial therapy within the CLL1320, CLL1411 or CLL17 trial will be analysed from first-line treatment, and OS, PFS and TTNT will also be analysed from second-line treatment.

Exploratory objectives:

Blood samples from all patients will be collected within routine clinical surveillance no more than once a year, to allow for exploratory analyses such as measurable residual disease (MRD) and other biomarkers.

Rationale for exploratory objectives:

The collection of blood samples, though seemingly interventional, can be scientifically justified since the collection aligns with routine clinical practice (during follow up in clinical routine, blood samples are required for each follow-up visit to assess the status of the disease). Because blood sampling is part of each routine visit, the blood samples drawn and collected for this study pose minimal physical and psychological risk to participants. Without the introduction of therapeutic or diagnostic interventions, analysis of blood samples may enable the identification of biomarkers that can help understand disease mechanisms, predict outcomes, or identify patient subgroups. The integration of blood sample data into an observational study bridges the gap between clinical observations and basic research. This can uncover molecular insights that drive innovation without altering the study's observational nature.

To maintain the integrity of the observational design, study participants will be fully informed about the purpose, use, and risks of blood sample collection. It will be explained in the patient informed consent form, that the consent to blood sampling is optional. No additional visit and no additional venal puncture will be required. By ensuring ethical and practical considerations, the study will maintain its observational nature while enabling valuable translational and clinical insights.

ELIGIBILITY:
Inclusion Criteria:

* • Subjects must voluntarily sign and date an informed consent, ap-proved by an independent ethics committee (IEC)/institutional review board (IRB)

  * Documented diagnosis of CLL at time point of inclusion in a first-line study of the GCLLSG (development of RT is not an exclusion criterion)
  * First-line treatment was administered within one of these first-line studies of the GCLLSG (CLL13, CLL14, or CLL17).
  * Subsequent therapy lines were either documented during the participa-tion in a first-line study of the GCLLSG or patient consented to have the subsequent therapy lines documented within this observational trial.
  * Subjects are willing and able to comply with procedures required in this protocol.

Exclusion Criteria:

* • Patients without participation in one of the first-line studies of the GCLLSG (CLL13, CLL14, CLL17)

  * Subjects with legal incapacity
  * Subjects who are institutionalized by regulatory or court order
  * Subjects who are in dependence to the sponsor or the investigator

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This observational trial will enrol patients who received first-line treatment in either CLL13, CLL14, or CLL17 trial. On ground of feasibility the sample size is estimat-ed at 1800-2000 patients in total. No formal sample size calculation has been performed.. The study population is defined as all patients who received first-line treatment in CLL13, CLL14, or CLL17 trial, regardless of whether they received any subse-quent lines of CLL therapy or not.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-08-01 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Each patient will be followed until death or end of study, whatever occurs first, i.e. 60 months from start nof enrolment.
  This observational trial is designed to investigate long-term survival with regard to the primary endpoint overall survival (OS) after start of first-line treatment.

CONTACTS AND LOCATIONS:
Overall Officials: BArbara F. Eichhorst, MD, Study Chair — Uniklinik Köln
Locations (1):
- University Hospital Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: Undecided